CLINICAL TRIAL: NCT04138264
Title: Opioid Consumption After Orthopaedic Surgery: Prospective Randomized Trial on the Effects of Pre-Operative Counseling
Brief Title: Opioid Counseling Following Orthopaedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ilyas2019
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peroperative counseling (Active Comparator)
  Interventions: Other: Preoperative opioid counseling
- No preoperative counseling (No Intervention)

INTERVENTIONS:
Other: Preoperative opioid counseling — preoperative counseling consists of education with a brief multi-media presentation in the preoperative area on the day of surgery using a handheld tablet. The message of the preoperative counseling consisted of: 1) Background on the opioid epidemic including basic facts and consequences, 2) Description of risk factors for opioid abuse and how to consume opioids safely, 3) Information on the specific opioid the patient was prescribed and the anticipated amount and duration of use postoperatively, 4) Encouraging the use of non-opioid therapy prior to taking the prescribed opioids or quickly transitioning to non-opioid medications postoperatively, and 5) Contact information and instructions to call if the patient experienced any adverse events and/or if additional pain medication is needed.
  Arms: Peroperative counseling

SUMMARY:
Postoperative pain management and opioid consumption following outpatient orthopaedic surgery may be influenced by a number of variables including knowledge of safe opioid use. A prospective randomized study is designed to understand the effect of preoperative opioid counseling on postoperative opioid consumption and the typical opioid consumption patterns following common outpatient orthopaedic surgeries. The hypothesis was that patients who received preoperative opioid counseling will consume less postoperative opioid medication and experience greater satisfaction with pain management.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing shoulder, elbow, wrist, knee, foot, and/or ankle surgery

Exclusion Criteria:

* male of female less than 18 years old
* patients schedule to undergo inpatient procedures
* patients undergoing surgeries distal to the wrist
* patients undergoing surgeries under local anesthesia only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Number of pills consumed | Up to 6 weeks
  Patients asked to keep daily diary which includes number of pills consumed during the post-operative period

SECONDARY OUTCOMES:
Morphine equivalents (MEQ) | Up to 6 weeks
  MEQs is a standardized method of comparing different types of pain medication with a gold-standard. All pain medication can be converted to MEQs
Visual Analog Scale (pain) Pain | Up to 6 weeks
  Pain as reported by patients on a daily basis via diaries
Patient satisfaction with pain management: 5 point Likert Scale | Up to 6 weeks
  Satisfaction with pain management as reported daily by patients using a 5 point Likert Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States